CLINICAL TRIAL: NCT01011842
Title: Comparison of Intrafraction Motion in Patients With Head and Neck Cancer Using Real-Time kV Imaging vs. Real-Time 3D Patient Surface Tracking
Brief Title: Real-Time kV Imaging vs. Real-Time 3D Patient Surface Tracking for Head & Neck Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Principal Investigator, Quynh-Thu Le, Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-16791; SU-09082009-3800 (Other: Stanford University); ENT0028 (Other: OnCore)
Record Dates: First submitted 2009-11-09; First posted 2009-11-11 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Radiotherapy; Radiation; Radiotherapy, Image-Guided

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- radiation therapy arm (Experimental)
  Interventions: Procedure: Radiotherapy; Procedure: Align RT

INTERVENTIONS:
Procedure: Radiotherapy — Standard of care
  Other Names: Radiation therapy; radiation oncology
Procedure: Align RT — Standard of care
  Other Names: Image-Guided Radiation Therapy

SUMMARY:
To determine if a new optical system that can track a patient's movement during treatment can be used to measure motion and allow for motion adjustments in order to decrease the amount of healthy tissue that receives radiation without limiting our ability to cure cancers using radiation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HNC undergoing radiation therapy at Stanford University
* Age >= 18 years old
* Radiation course >= 4 weeks duration
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Factors such as claustrophobia inhibiting use of thermoplastic mask immobilization device.
* Patients who are pregnant or nursing, which preclude them from undergoing active radiation treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
We are measuring how much a patient moves during treatment. | This information will be available immediately have the patient is treated.

CONTACTS AND LOCATIONS:
Overall Officials: Quynh-Thu Le, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No